CLINICAL TRIAL: NCT04786457
Title: A Phase 1, Open-Label Clinical Trial With Dengue-1-Virus Live Virus Human Challenge (DENV-1-LVHC) Assessment of Healthy U.S. Adults Previously Primed With Tetravalent Dengue Virus Purified Inactivated Vaccine (TDEN-PIV) and Boosted With Tetravalent Dengue Virus Live Attenuated Vaccine Formulation (TDEN LAV)
Brief Title: ADVP005; Dengue CVD 12000 - Dengue-1-Virus Live Virus Human Challenge (DENV-1-LVHC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: United States Army Medical Materiel Development Activity (U.S. Federal Agency); Medical Technology Enterprise Consortium (MTEC) (Unknown)
Responsible Party: Principal Investigator, Kirsten Lyke, Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00088798
Record Dates: First submitted 2020-11-24; First posted 2021-03-08 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dengue 1 Live Virus Human Challenge (DENV-1-LVHC) (Experimental): open-label injection of DENV-1-LVHC to 15-20 adults who were previously vaccinated and 5 adults who have never received a dengue vaccination
  Interventions: Biological: Dengue 1 Live Virus Human Challenge (DENV-1-LVHC)

INTERVENTIONS:
Biological: Dengue 1 Live Virus Human Challenge (DENV-1-LVHC) — one subcutaneous injection of Dengue 1 Live Virus Human Challenge (DENV-1-LVHC) at 0.5 mL of 6.5 x 10^3 PFU/mL

SUMMARY:
The purpose of this research study is to test the protection of volunteers previously vaccinated with Tetravalent Dengue Virus (TDEN) Purified Inactivated Vaccine (PIV) with alum and boosted with TDEN live attenuated vaccine (LAV) formulation against a weakened form of an experimental dengue virus challenge. The Investigators will also include people that have not received the study vaccine. The Investigators are collecting information about how the vaccine protects against a dengue virus challenge as well as adding to knowledge about the safety of the challenge.

DETAILED DESCRIPTION:
The purpose of this research study is to test the protection of volunteers previously vaccinated with Tetravalent Dengue Virus (TDEN) Purified Inactivated Vaccine (PIV) with alum and boosted with TDEN live attenuated vaccine (LAV) formulation against a weakened form of an experimental dengue virus challenge. The Investigators will also include people that have not received the study vaccine. The Investigators are collecting information about how the vaccine protects against a dengue virus challenge as well as adding to knowledge about the safety of the challenge. The information will help Investigators develop vaccines to protect people from dengue. Participation is voluntary. The duration of participation will last for 180 days (six months). After participants are exposed to the weakened dengue virus, the Investigators will follow them closely to measure their symptoms. Like the flu, participants might expect to have a headache, rash, body aches, fever and chills or they may experience no symptoms whatsoever. If a participant does develops symptoms, the Investigators will monitor him/her closely in a local hotel or a wing of our hospital to ensure safety and to treat symptoms if they occur. Participants will be compensated for their time.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or non-pregnant, non-breastfeeding female between 18 and 50 years of age (inclusive) at the time of consent.
* 2. Tetravalent dengue antibody response at 28 days following final vaccination for vaccinated groups of volunteers.
* 3. Volunteers must be able and willing to provide written informed consent.
* 4. Volunteers must be healthy as established by medical history and clinical examination at study entry.
* 5. Volunteers must pass a comprehension test and be able to comply with all study requirements.
* 6. Female volunteers of non-childbearing potential (non-childbearing potential is defined as having had one of the following: a tubal ligation at least 3 months prior to enrollment, a hysterectomy, an oophorectomy, or is post-menopausal).
* 7. Female volunteers of childbearing potential may be enrolled in the study, if all of the following apply:
* Practiced adequate contraception (see Definition of Terms, section 5.4.2.3.) for 30 days prior to challenge
* Has a negative urine pregnancy test on the day of DHIM
* Agrees to continue adequate contraception until two months after completion of the DHIM
* 8. Provide consent for release of medical history records from primary care physician, college or university medical center, urgent care, or emergency room visit

Exclusion Criteria:

* 1. Planned travel during the study period (180 days) which would interfere with the ability to complete all study visits
* 2. Recent (in the past 4 weeks) travel to any dengue endemic area. These potential volunteers may be eligible for enrollment a minimum of 4 weeks later
* 3. Volunteer seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV)
* 4. Unvaccinated volunteers positive for antibodies to flaviviruses (FV) to include dengue virus, West Nile virus, Yellow Fever virus, Zika virus, and Japanese encephalitis virus.
* 5. Any history of FV infection or FV vaccination except for participation in the ADVP003 or ADVP004 dengue vaccination studies; during the study period (Note: Late time point serology from the trials can be tested concomitant to screening serology to clarify if incident FV infection has occurred between vaccination and challenge)
* 6. Medical history of, or current, diabetes, chronic obstructive pulmonary disease, peptic ulcer disease, coronary artery disease, cardiac arrhythmia, cardiomyopathy, pericarditis, or auto-immune disease
* 7. Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* 8. History of Guillain-Barré syndrome (GBS)
* 9. History of bipolar disorder, schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition, which in the opinion of the investigator prevents the volunteer from participating in the study
* 10. Safety laboratory test results at screening that are deemed clinically significant or more than Grade 1 deviation from normal with the exception of PT/PTT, fibrinogen decrease, ALT/AST increase (<1.1 x ULN acceptable), platelet decrease which will be exclusionary at Grade 1 or higher
* 11. Significant screening physical examination abnormalities at the discretion of the investigator, including a BMI > 35 kg/m2
* 12. Women who intend to become pregnant or men who intend to father a child during the study period (approximately 6 months)
* 13. Female: pregnant, lactating or history of heavy menstrual bleeding menstrual periods lasting consistently and regularly longer than 6 days, or consistently and regularly requiring 5 or more pads or tampons per day, and volunteer to the opinion and review of the investigator.
* 14. Female volunteers using an intrauterine device (IUD) or Mirena®
* 15. Female volunteers with a history of clinically significant fibroids or uterine polyps, endometriosis, dysmenorrhea, adenomyosis, and uterine scarring (e.g. after D&C), unless treated, with no active clinically significant disease
* 16. Allergy (hives, shortness of breath, swelling of the lips or throat), or hospitalization related to a previous vaccination, anaphylaxis of unknown etiology, or allergy to specific medications/animals for which antigens may be in the virus preparations to include: Shellfish allergy, Fetal Bovine Serum, L-Glutamine, Neomycin and Streptomycin
* 17. Recent blood donation within prior 56 days of inoculation or planning to donate blood in the one 1 year following inoculation with dengue virus
* 18. Receipt of blood products or antibodies within 90 days of inoculation or during the study period
* 19. Any personal beliefs that bar the administration of blood products, transfusions, or serum albumin
* 20. Participation in the 4 weeks preceding inoculation, or planned participation during the present trial period, in another clinical trial investigating a vaccine except for participation in the ADVP003 or ADVP004 study, drug, medical device, or medical procedure
* 21. Planned administration of a licensed or study vaccine not planned in the study protocol during the period starting 30 days prior to the DHIM for a live vaccine or 14 days prior to DHIM for inactivated vaccines and extending until 56 days after study completion
* 22. Planned or current administration of an HMG-CoA reductase inhibitor (i.e., lovastatin, simvastatin, atorvastatin, etc.)
* 23. Currently taking methadone or suboxone
* 24. Currently regularly taking anti-coagulant medication, aspirin or non-steroidal anti-inflammatory drugs (NSAIDs)
* 25. Chronic migraine headaches, defined as more than 15 headache days per month over a 3-month period of which more than 8 are migraines, in the absence of medication over use
* 26. Chronic or recent acute medical condition that, in the opinion of the investigator, impacts volunteer safety.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lyke KE, Chua JV, Koren M, Friberg H, Gromowski GD, Rapaka RR, Waickman AT, Joshi S, Strauss K, McCracken MK, Gutierrez-Barbosa H, Shrestha B, Culbertson C, Bernal P, De La Barrera RA, Currier JR, Jarman RG, Edelman R. Efficacy and immunogenicity following dengue virus-1 human challenge after a tetravalent prime-boost dengue vaccine regimen: an open-label, phase 1 trial. Lancet Infect Dis. 2024 Aug;24(8):896-908. doi: 10.1016/S1473-3099(24)00100-2. Epub 2024 Apr 25. PMID 38679035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 volunteers assessed - 6 ineligible (lab results n = 4, abnormal physical findings n = 1, Other n = 1), Decline participation n = 2
Groups:
- Vaccinees: Previously vaccinated with: Tetravalent Dengue Virus (TDEN) Purified Inactivated Vaccine (PIV) with Alum adjuvant prime and boosted with tetravalent live attenuated Dengue virus vaccine
- Controls: Not previously vaccinated with tetravalent dengue vaccine
Period: Overall Study
Arm/Group | Vaccinees | Controls
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vaccinee: Recipient of tetravalent dengue prime boost vaccine
- Control: Dengue and flavivirus naive
- Total: Total of all reporting groups
Arm/Group | Vaccinee | Control | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 32.5 [26 to 41] | 40.7 [34 to 47] | 36.6 [26 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 1 | 2 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Injection Site Adverse Events
Description: Number of Participants with Solicited Injection Site Erythema - solicited injection site adverse event until 7 days post virus inoculation
Time Frame: Days 2, 4, 5, 6, and 7
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 6 | 4
Participants | 0 | 1

2. Primary Outcome: Number of Participants With Unsolicited Injection Site Adverse Events
Description: Number of Participants with Injection site pain - unsolicited injection site adverse events until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: Days 2, 4, 5-16, 28 (until 28 days post virus inoculation or 7 days post hospitalization, whichever is later, up to a maximum of 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 6 | 4
Participants | 0 | 1

3. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events
Description: Number of participants with solicited systemic adverse events until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: Days 2, 4-16, 19, 22, 25, and 28 (until 28 days post virus inoculation or 7 days post hospitalization, whichever is later, up to a maximum of 28 days)
Measure: Number; unit: participants
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 5 | 4
participants
  Fever | 4 | 2
  Abdominal Pain | 2 | 2
  Eye pain / Headache | 5 | 4
  Muscle Pain | 4 | 4
  Joint or Bone Pain | 3 | 2
  Fatigue | 4 | 4
  Nausea or Vomiting | 3 | 1
  Rash | 3 | 4

4. Primary Outcome: Number of Participants With Incidence of Abnormal Laboratory Measurements
Description: Number of participants with incidence of abnormal laboratory measurements until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 5 | 4
participants
  Leukopenia | 4 | 4
  Thrombocytopenia | 0 | 1
  AST | 4 | 3
  ALT | 4 | 3
  Fibrinogen | 1 | 0

5. Primary Outcome: Dengue-Related Illness Index
Description: Scales:
  Clinical Symptoms: None=0, Mild=1, Moderate=2, Severe=3 (Min Score=0, Max=3) Laboratory Abnormalities: None=0, Mild=1, Moderate=2, Severe=3 based on modified FDA CBER laboratory scale (per protocol) (Min=0, Max=3) Symptoms (Clinical symptoms or Laboratory Abnormalities) duration: 1 point/day (Day 1-16) (Min=0, Max=16) Subscale A (Symptom Duration): 1 point/day (Day 1-16) across 10 Clinical/Laboratory findings (Min = 0, Max = 160) Subscale B (Symptom # per day): 1 point/ Clinical/Laboratory finding (n=10) per day across 16 days Min=0, Max=160 Subscale C (Max Severity Score/day): None=0, Mild=1, Moderate=2, Severe=3 across 16 days: Min=0, Max=48 Total Range in DII score (total scale) which equates to subscale (A + B + C)/3: Min=0, Max=122.7
  https://doi.org/10.1016/s1473-3099(24)00100-2.
Time Frame: Days 1-16
Population: only people with dengue were assessed (n=9).
Measure: Mean (Full Range); unit: Dengue-Related Illness Index Score
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 5 | 4
Dengue-Related Illness Index Score | 19.4 [15.7 to 22] | 23.1 [21 to 26.7]

6. Primary Outcome: Number of Participants With Unsolicited Systemic Adverse Events
Description: Number of participants with unsolicited systemic adverse events until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 6 | 4
participants
  Gastrointestinal Upset | 0 | 1
  Generalized Muscle Pain | 0 | 1
  Headache | 0 | 1
  Shoulder Pain - Left | 1 | 0
  Lower Back Pain | 0 | 1

7. Primary Outcome: Number of Participants With Short-Term SAEs
Description: Number of participants with SAEs until 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

8. Primary Outcome: Number of Participants With Long-Term SAEs
Description: Number of participants with SAEs until 6 months post virus inoculation
Time Frame: Days 2-180
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

9. Primary Outcome: Number of Participants With Persistent Fever
Description: Number of participants with persistent fever defined as greater than or equal to 38°C (100.4° F) measured at least 2 times at least 4 hours apart
Time Frame: Days 2-28
Population: Per protocol analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinees | Controls
Number analyzed (Participants) | 6 | 4
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: Local injection site adverse events were collected through day 7 post challenge. Solicited, unsolicited, and solicited lab adverse events were collected through Day 28. SAEs were also collected through 6-months post inoculation.
Description: Daily AEs were assessed.
Arm/Group | Vaccinees | Controls
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 5/6 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccinees (N=6) | Controls (N=4)
Injection Site Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Injection Site Pain (General disorders) | 0 | 1
Fever (Immune system disorders) | 4 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Eye Pain / Headache (General disorders) | 5 | 4
Muscle Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Joint or Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Fatigue (Immune system disorders) | 4 | 4
Nausea or Vomiting (Gastrointestinal disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT04786457/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04786457/SAP_001.pdf